CLINICAL TRIAL: NCT06241313
Title: Randomized, Double-blind, Placebo-Controlled, Multiple-Attack Study With an Open-Label Extension to Evaluate the Efficacy, Safety, Tolerability, and the Consistency of Effect of Atogepant for the Acute Treatment of Migraine (ECLIPSE)
Brief Title: Study of Oral Atogepant Tablets to Assess Safety and Efficacy in Adult Participants With Migraine
Acronym: ATO ACUTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-305; 2023-506029-12-00 (Other: EU CT)
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Migraine; Atogepant; ECLIPSE; Qulipta; Aquipta
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sequence 1 (Placebo Comparator): Participants will receive both atogepant and placebo to treat qualifying migraines.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant
- Sequence 2 (Experimental): Participants will receive both atogepant and placebo to treat qualifying migraines.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant
- Sequence 3 (Experimental): Participants will receive both atogepant and placebo to treat qualifying migraines.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant
- Sequence 4 (Experimental): Participants will receive both atogepant and placebo to treat qualifying migraines.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: Qulipta; Aquipta
Drug: Placebo for Atogepant — Oral Tablet

SUMMARY:
A migraine attack is a moderate or severe headache that usually occurs on one side of the head and is often accompanied by throbbing, sensitivity to light, sensitivity to sound, nausea, or other symptoms. The main goal of the study is to see if atogepant is effective, safe, and well-tolerated in treating migraine attacks quickly.

Atogepant is a medicine currently approved for the preventive treatment of migraine in adults and has been shown to be effective and well tolerated when taken daily to prevent migraine attacks. This study includes double-blind phase means that neither the participants nor the study doctors know who is given which study treatment (atogepant or placebo) followed by an open-label phase meaning that both participants and study doctors know which study treatment is given. All participants will receive atogepant during the open-label part of the study. This study will include 1300 participants aged 18-75 years with a history of migraine at approximately 160 sites across the world.

All participants will receive both atogepant and placebo to treat qualifying migraines. At the start of the study, participants will be randomized to 1 of 4 dosing sequences to determine when they will receive atogepant and when they will receive placebo during the study. After treating 4 qualifying migraine attacks, participants will receive open-label atogepant for any additional migraine attacks they have until the end of the study (Week 24).

There may be a bigger responsibility for participants in this study than there would be in participants receiving standard of care treatment. participants will attend regular visits during the study at a hospital or clinic, as well as telephone visits, and the effects of treatment will be checked by completion of questionnaires in an electronic diary, medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine (with or without aura) according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) for >= 12 months prior to Visit 1/Screening.
* History of 2 to 8 migraine attacks of moderate to severe headache pain in each of the 3 months prior to Visit 1/Screening per investigator judgment.
* Migraine onset before the age of 50.
* History of migraines lasting between 4 and 72 hours when untreated or treated unsuccessfully and migraine episodes separated by at least 48 hours of headache pain freedom.

Exclusion Criteria:

* History of an average of 15 or more headache days per month in the 6 months prior to Visit 1/Screening per the investigator's judgment, or a current diagnosis of chronic migraine as defined by ICHD-3.
* Require hospital/emergency room treatment for migraine attacks on 3 or more occasions within 6 months prior to Visit 1/Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Pain Freedom at 2 Hours After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Pain freedom is defined as a reduction in headache severity from moderate/severe at baseline (predose) to no pain.

SECONDARY OUTCOMES:
Percentage of Participants With Absence of Most Bothersome Migraine-associated Symptom (MBS) at 2 Hours After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Percentage of Participants With Absence of Most Bothersome Migraine-associated Symptom (MBS) will be assessed.
Percentage of Participants Achieving Pain Relief at 2 Hours After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Pain relief is defined as the reduction of a moderate/severe migraine headache at baseline [predose] to a mild headache or to no headache.
Percentage of Participants Achieving Sustained Pain Relief From 2 to 24 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Sustained pain relief is defined as pain relief at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a moderate/severe headache from 2 to 24 hours.
Percentage of Participants Achieving Sustained Pain Relief From 2 to 48 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Sustained pain relief is defined as pain relief at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a moderate/severe headache from 2 to 24 hours.
Percentage of Participants With Use of Rescue Medication Within 24 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Percentage of participants with use of rescue medication within 24 hours after the DB dose for the first attack will be assessed.
Percentage of Participants With Ability to Function Normally at 2 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Percentage of participants with ability to function normally at 2 hours after the DB dose for the first attack will be assessed.
Percentage of Participants Achieving Sustained Pain Freedom From 2 to 24 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Sustained pain freedom is defined as pain freedom at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a mild/moderate/severe headache from 2 to 24 hours.
Percentage of Participants Achieving Sustained Pain Freedom From 2 to 48 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Sustained pain freedom is defined as pain freedom at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a mild/moderate/severe headache from 2 to 24 hours.
Percentage of Participants With Absence of Photophobia at 2 Hours After the DB Dose for the First Attack | Approximately 16 Weeks
  Photophobia is defined as sensitivity to light.
Percentage of Participants With Absence of Phonophobia at 2 Hours After the DB Dose for the First Attack | Approximately 16 Weeks
  Phonophobia is defined as sensitivity to sound.
Percentage of Participants Achieving Pain Freedom at 8 Hours After the DB Dose for the First Attack | Approximately 16 Weeks
  Pain freedom is defined as a reduction in headache severity from moderate/severe at baseline (predose) to no pain.
Percentage of Participants With Ability to Function Normally at 8 Hours After DB Dose for the First Attack | Approximately 16 Weeks
  Percentage of participants with ability to function normally at 8 hours after the DB dose for the first attack will be assessed.
Percentage of Participants Achieving Pain Relief at 1 Hour After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Pain relief is defined as the reduction of a moderate/severe migraine headache at baseline [predose] to a mild headache or to no headache.
Percentage of Participants With Absence of Nausea at 2 Hours After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Percentage of participants with absence of nausea at 2 hours after the DB dose for the first attack.
Percentage of Participants Achieving Pain Relief at 30 Minutes After the Double-Blind (DB) Dose for the First Attack | Approximately 16 Weeks
  Pain relief is defined as the reduction of a moderate/severe migraine headache at baseline [predose] to a mild headache or to no headache.
Percentage of Participants With Ability to Function Normally at 1 Hour After DB Dose for the First Attack | Approximately 16 Weeks
  Percentage of participants with ability to function normally at 1 hour after the DB dose for the first attack will be assessed.
Percentage of Participants Achieving Pain Freedom at 2 Hours After Receiving DB Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Pain freedom is defined as a reduction in headache severity from moderate/severe at baseline (predose) to no pain.
Percentage of Participants Achieving Pain Relief at 2 Hours After Receiving Double-Blind (DB) Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Pain relief is defined as the reduction of a moderate/severe migraine headache at baseline [predose] to a mild headache or to no headache.
Percentage of Participants Achieving Sustained Pain Freedom From 2 to 24 Hours After Receiving DB Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Sustained pain freedom is defined as pain freedom at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a mild/moderate/severe headache from 2 to 24 hours.
Percentage of Participants Achieving Sustained Pain Freedom From 2 to 48 Hours After Receiving DB Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Sustained pain freedom is defined as pain freedom at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a mild/moderate/severe headache from 2 to 24 hours.
Percentage of Participants Achieving Sustained Pain Relief From 2 to 24 Hours After Receiving DB Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Sustained pain relief is defined as pain relief at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a moderate/severe headache from 2 to 24 hours.
Percentage of Participants Achieving Sustained Pain Relief From 2 to 48 Hours After Receiving DB Atogepant for at least 2 out of 3 Attacks | Approximately 16 Weeks
  Sustained pain relief is defined as pain relief at 2 hours after the DB dose with no administration of rescue medication and no occurrence of a moderate/severe headache from 2 to 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (149):
- Belgium (8):
  - Universitair Ziekenhuis Antwerpen /ID# 257582, Edegem, Antwerpen
  - Universitair Ziekenhuis Brussel /ID# 257584, Jette, Brussels Capital
  - Jessa Ziekenhuis /ID# 257578, Hasselt, Limburg
  - AZ Sint-Jan Brugge /ID# 257585, Bruges, West-Vlaanderen
  - AZ Groeninge /ID# 257586, Kortrijk
  - H.-Hartziekenhuis Lier /ID# 257577, Lier
  - CHR de la Citadelle /ID# 257587, Liège
  - Cabinet Prive Dr Sava /ID# 257581, Saint-Nicolas
- China (35):
  - The first affiliated hospital of bengbu medical college /ID# 258758, Bengbu, Anhui
  - Beijing Friendship Hospital /ID# 258830, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University /ID# 258510, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 259573, Beijing, Beijing Municipality
  - Chinese PLA General Hospital /ID# 257540, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 258672, Xicheng District, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 259575, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University /ID# 259576, Xiamen, Fujian
  - Lanzhou University Second Hospital /ID# 259667, Lanzhou, Gansu
  - Guangzhou First People's Hospital /ID# 258656, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University /ID# 258638, Guangzhou, Guangdong
  - The University Of Hong Kong - Shenzhen Hospital /ID# 258462, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University /ID# 259536, Guiyang, Guizhou
  - Hainan General Hospital /ID# 259548, Haikou, Hainan
  - Hebei General Hospital /ID# 258583, Shijiazhuang, Hebei
  - Zhengzhou People's Hospital /ID# 258670, Zhengzhou, Henan
  - The Second Xiangya Hospital Of Central South University /ID# 260623, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University /ID# 258787, Changsha, Hunan
  - Zhuzhou Central Hospital /ID# 260076, Zhuzhou, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University /ID# 258648, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University /ID# 259551, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 258783, Suzhou, Jiangsu
  - Jiangxi Pingxiang Peoples Hospital /ID# 258652, Pingxiang, Jiangxi
  - The First Hospital of Jilin University /ID# 259585, Changchun, Jilin
  - The Second hospital of Jilin university /ID# 258556, Changchun, Jilin
  - General Hospital of Northern Theater Command /ID# 259556, Shenyang, Liaoning
  - Shaanxi Provincial PeopleS Hospital /ID# 259529, Xi'an, Shaanxi
  - Second Hospital of Shanxi Medical University /ID# 259669, Taiyuan, Shanxi
  - West China Hospital, Sichuan University /ID# 258664, Chengdu, Sichuan
  - Tianjin Medical University General Hospital /ID# 259513, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital /ID# 258625, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 258860, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 258939, Wenzhou, Zhejiang
  - Baotou Central Hospital /ID# 258786, Baotou
  - The first people's Hospital Affiliated to Shanghai Jiaotong University /ID# 259554, Shanghai
- Czechia (11):
  - CCR Ostrava, s.r.o. /ID# 257743, Ostrava, Ostrava-mesto
  - Fakultni Nemocnice Ostrava /ID# 259023, Ostrava, Ostrava-mesto
  - Praglandia /ID# 257667, Prague, Praha 5
  - NeuroHK s.r.o. /ID# 257671, Hradec Králové
  - Clintrial s.r.o. /ID# 257663, Prague
  - DADO MEDICAL s.r.o. /ID# 257672, Prague
  - Axon Clinical, s.r.o. /ID# 259024, Prague
  - Fakultni Thomayerova nemocnice /ID# 259021, Prague
  - FORBELI s.r.o. /ID# 259019, Prague
  - INEP medical s.r.o. /ID# 257669, Prague
  - Vestra Clinics s.r.o. /ID# 259022, Rychnov nad Kněžnou
- Germany (10):
  - Neuropraxis Muenchen Sued /ID# 258077, Unterhaching, Bavaria
  - Kopfschmerzzentrum - Frankfurt /ID# 258019, Frankfurt am Main, Hesse
  - Studienzentrum Nord-West /ID# 258024, Westerstede, Lower Saxony
  - Universitaetsklinikum Duesseldorf /ID# 258078, Düsseldorf, North Rhine-Westphalia
  - Ambenet Hausarztpraxis /ID# 258075, Leipzig, Saxony
  - Schmerzklinik Kiel /ID# 258005, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 258076, Berlin
  - Universitaetsklinikum Essen /ID# 258023, Essen
  - Vitos Orthopaedische Klinik Kassel gemeinnuetzige GmbH /ID# 258008, Kassel
  - Velocity Clinical Research /ID# 258020, Wiesbaden
- Hungary (6):
  - Jávorszky Ödön Kórház /ID# 258969, Vác, Pest County
  - Cortex Study Center /ID# 259032, Budapest
  - Semmelweis Egyetem /ID# 258546, Budapest
  - Semmelweis Egyetem /ID# 258800, Budapest
  - UNO Medical Trials /ID# 259186, Budapest
  - S-Medicon Kft /ID# 258547, Budapest
- Italy (11):
  - Istituto Neurologico Mediterraneo Neuromed /ID# 258593, Pozzilli, Isernia
  - ASL 1 Abruzzo - Ospedale SS. Filippo and Nicola /ID# 258590, Avezzano, L Aquila
  - IRCCS Ospedale San Raffaele /ID# 258592, Milan, Milano
  - Istituto Auxologico Italiano - Irccs /ID# 258623, Milan, Milano
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 258591, Turin, Piedmont
  - Univ. of Bologna-IRCCS-Istituto delle Scienze Neurologiche /ID# 261089, Bologna
  - ASST degli Spedali Civili di Brescia /ID# 258594, Brescia
  - ICOT Istituto Marco Pasquali /ID# 258621, Latina
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS /ID# 258589, Pavia
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 258588, Roma
  - Ospedale San Paolo - ASL2 /ID# 258622, Savona
- Japan (11):
  - Tokyo Dental College Ichikawa General Hospital /ID# 259570, Ichikawa-shi, Chiba
  - Ikeda Neurosurgical Clinic /ID# 259085, Kasuga-shi, Fukuoka
  - Higashi Sapporo Neurology And Neurosurgery Clinic /ID# 262708, Sapporo, Hokkaido
  - Umenotsuji Clinic /ID# 258717, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 258862, Sendai, Miyagi
  - Tominaga Clinic - Osaka /ID# 258553, Osaka, Osaka
  - Usuda Clinic Of Internal Medicine /ID# 260422, Setagaya-ku, Tokyo
  - Tokyo Headache Clinic /ID# 258534, Shibuya-ku, Tokyo
  - Nagaseki Headache Clinic /ID# 259214, Kai, Yamanashi
  - DOI Internal Medicine-Neurology Clinic /ID# 259009, Hiroshima
  - Tatsuoka Neurology Clinic /ID# 258771, Kyoto
- Poland (10):
  - Solumed Centrum Medyczne /ID# 258288, Poznan, Greater Poland Voivodeship
  - Clinical Research Center Medic-R /ID# 258268, Poznan, Greater Poland Voivodeship
  - Vitamed Galaj i Cichomski Sp.j. /ID# 258278, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Athleticomed Sp. z o.o /ID# 258253, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Linden Sp. z o.o. sp.k. /ID# 258283, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska Jedynak /ID# 258248, Oświęcim, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 258281, Lublin, Lublin Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 258250, Gdansk, Pomeranian Voivodeship
  - Silmedic Sp. z o.o. /ID# 258249, Katowice, Silesian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 258287, Wroclaw
- Portugal (6):
  - Unidade Local de Saude do Alto Ave, EPE /ID# 257986, Guimarães, Braga District
  - Unidade Local de Saude de Almada-Seixal, EPE /ID# 257987, Almada, Setúbal District
  - Hospital da Luz Lisboa /ID# 257983, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 257989, Lisbon
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 258140, Porto
  - Unidade Local de Saude da Arrabida, EPE /ID# 258139, Setúbal
- Slovakia (6):
  - Univerzitna nemocnica - Nemocnica svateho Michala a.s. /ID# 257909, Bratislava, Bratislava Region
  - Poliklinika Bezrucova (Cliniq s.r.o.) /ID# 257961, Bratislava, Bratislava Region
  - University Hospital Bratislava - Hospital ak. L. Derera /ID# 257947, Bratislava, Bratislava Region
  - Neurologicka a algeziologicka ambulancia, SANERA /ID# 259176, Prešov, Presov
  - MUDr. Beata Dupejova neurologicka ambulancia s.r.o. /ID# 257901, Banská Bystrica
  - Liptovska nemocnica s poliklinikou MUDr. Ivana Stodolu Liptovsky Mikulas /ID# 258315, Liptovský Mikuláš, Žilina Region
- South Korea (6):
  - Hallym University Dongtan Sacred Heart Hospital /ID# 257999, Hwaseong, Gyeonggido
  - Chonnam National University Hospital /ID# 259154, Gwangju, Jeonranamdo
  - Nowon Eulji Medical Center, Eulji University /ID# 258000, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 258002, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 258001, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 257998, Seoul
- Spain (8):
  - Hospital Universitario Marques de Valdecilla /ID# 257658, Santander, Cantabria
  - Clinica Universidad de Navarra - Pamplona /ID# 257656, Pamplona, Navarre
  - Hospital Universitario Vall de Hebron /ID# 257652, Barcelona
  - Hospital Universitario La Paz /ID# 257654, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 257657, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 257655, Valencia
  - Hospital Clinico Universitario de Valladolid /ID# 257653, Valladolid
  - Hospital Clinico Universitario Lozano Blesa /ID# 257661, Zaragoza
- Sweden (5):
  - Skaneuro Privatmottagning /ID# 258833, Lund, Skåne County
  - Karolinska Universitetssjukhuset - Huddinge /ID# 258837, Huddinge, Stockholm County
  - Neurology Clinic /ID# 258835, Stockholm, Stockholm County
  - CTC EbbePark Linkoping /ID# 261170, Linköping
  - Optimuskliniken /ID# 258834, Upplands Vasby
- Taiwan (5):
  - Kuang-Tien General Hospital /ID# 258063, Taichung, Taichung
  - Taipei Veterans General Hospital /ID# 258062, Taipei City, Taipei
  - China Medical University Hospital /ID# 258417, Taichung
  - Tri-Service General Hospital /ID# 258064, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 259171, Taoyuan
- United Kingdom (11):
  - St Pancras Clinical Research /ID# 277704, Chester, Cheshire
  - North Coast Medical Ltd - Newquay Health Centre /ID# 260019, Newquay, Cornwall
  - Ashgate Medical Practice /ID# 258923, Chesterfield, Derbyshire
  - The Adam Practice /ID# 258190, Poole, Dorset
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde /ID# 259384, Glasgow, Lanarkshire
  - Re:Cognition Health Birmingham /ID# 258186, Birmingham
  - Re:Cognition Health Bristol /ID# 258187, Bristol
  - Re:Cognition Health - Guildford /ID# 258188, Guildford
  - St Pancras Clinical Research /ID# 258183, London
  - The University of Nottingham Health Service /ID# 259380, Nottingham
  - Primary Care Sheffield /ID# 259448, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-305